CLINICAL TRIAL: NCT07069608
Title: Cheers Health Restore Observational Study
Brief Title: Cheers Health Restore Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cheers Health (Industry)
Collaborators: Alethios, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1002
Record Dates: First submitted 2025-06-18; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Sleep; Alcohol Aftereffects; Recovery
Keywords: alcohol use; wellness
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Cheers Restore — Cheers Restore contains a formulation of antioxidants, electrolytes, and plant-based compounds designed to support physiological resilience and sleep recovery after alcohol consumption. This study is structured to evaluate Cheers Restore in a real-world setting without introducing investigational or therapeutic claims.

SUMMARY:
This observational cohort study, sponsored by Cheers Health and conducted by Principal Investigator Dr. Nirav Shah, aims to evaluate the potential role of Cheers Restore in supporting sleep quality, physiological recovery, and next-day well-being following alcohol consumption in healthy adults. Over a 6 week period, the study will utilize wearable devices and self-reported outcomes captured via the Alethios platform to assess real-world responses to use of Cheers Restore. Outcomes will be compared across three behavioral conditions: (1) alcohol consumption followed by Cheers Restore use, (2) alcohol-only nights without use of Cheers Restore, and (3) non-drinking nights.

DETAILED DESCRIPTION:
Alcohol consumption is known to reduce REM sleep, impair heart rate variability (HRV), and increase next-day fatigue, irritability, and cognitive disruption. Moderate alcohol intake can disrupt circadian rhythm and impair autonomic recovery. Prior research has shown dietary supplements containing amino acids, antioxidants, and electrolytes may support recovery, but few studies have assessed real-world behavioral patterns using digital health technology. Observational data from wearable devices and participant-reported outcomes can offer scalable, ecologically valid insights into how lifestyle products may mitigate alcohol-induced disruption.

Cheers Restore contains a formulation of antioxidants, electrolytes, and plant-based compounds designed to support physiological resilience and sleep recovery after alcohol consumption. This study is structured to evaluate Cheers Restore in a real-world setting without introducing investigational or therapeutic claims. By capturing participant-driven usage patterns and outcomes, the study enables ecological validation and supports responsible product communication aligned with DSHEA and FTC guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 years or older
* Regular alcohol consumers (defined as ≥1 drinking night per week)
* Ownership of and willingness to use a wearable device compatible with the Alethios platform (e.g., Fitbit, Apple Watch, Oura)
* Ability and willingness to log alcohol consumption, Cheers Restore usage, and complete daily and weekly surveys via smartphone or web
* Willingness to use Cheers Restore during the study period when consuming alcohol
* English-speaking, capable of understanding informed consent

Exclusion Criteria:

* AUDIT-C score above gender-specific thresholds for hazardous drinking (≥4 for men, ≥3 for women)
* History of alcohol use disorder or prior treatment for substance misuse
* Routine binge drinking (≥5 drinks/occasion for men, ≥4 for women)
* Use of confounding substances:
* THC (any form)
* Recreational drugs
* Prescription stimulants, sedatives, or sleep aids
* Diagnosed sleep or psychiatric conditions known to impair sleep quality (e.g., insomnia, obstructive sleep apnea, restless legs syndrome, narcolepsy, major depressive disorder, post-traumatic stress disorder, bipolar disorder, schizophrenia, attention deficit/hyperactivity disorder)
* Pregnancy or breastfeeding
* Anticipated travel or scheduling conflicts disrupting normal sleep/alcohol routines
* Inability to comply with platform-based data collection requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a decentralized, 6 week observational cohort study conducted via the Alethios platform with approximately 100 participants.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | 6 weeks
  Sleep quality, as measured by wearables such as Fitbit, Garmin and Oura rings (time spent in sleep stages, wakeup events, sleep onset).

SECONDARY OUTCOMES:
Alcohol Consumption Behavior | 6 weeks
  Alcohol consumption behavior, including quantity (number of standard drinks), frequency of alcohol consumption, and timing as measured by weekly surveys.
Heart Rate Variability | 6 weeks
  Heart Rate Variability during sleep as measured by wearable devices e.g. Garmin, Oura, Fitbit.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Cheers Restore Observational Study Landing Page and Eligibility Questionnaire — https://studies.alethios.com/cheers-restore-observational-study